CLINICAL TRIAL: NCT04954391
Title: Pulsed Radiofrequency of the Suprascapular, Axillary Nerve and Articular Branch of the Lateral Pectoral Nerve vs Pulsed Radiofrequency of the Suprascapular Nerve Only for Chronic Shoulder Pain. A Prospective Randomized Double-blind Study
Brief Title: Pulsed Radiofrequency One or Three Nerves for Chronic Shoulder Pain. A Prospective, Randomized, Double-blind Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Saint Petersburg State University, Russia (Other)
Responsible Party: Principal Investigator, Konstantin Truhin, anesthesiologist, Saint Petersburg State University, Russia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 06/21
Record Dates: First submitted 2021-06-20; First posted 2021-07-08 (Actual); Last update posted 2023-05-23 (Actual); Status verified 2023-05

CONDITIONS: Chronic Shoulder Pain
Keywords: chronic shoulder pain; pulsed radiofrequency; suprascapular nerve; axillary nerve; lateral pectoral nerve; shoulder arthroscopy; rotator cuff injury; adhesive capsulitis; subacromial impingement; glenohumeral arthrosis; acromioclavicular joint
MeSH Terms: conditions — Rotator Cuff Injuries; Bursitis; Shoulder Impingement Syndrome

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PRF one nerve (Active Comparator): Ultrasound guided PRF neuromodulation of suprascapular nerve and block axillary nerve, and articular branch of the lateral pectoral nerve with ropivacaine and dexamethasone
  Interventions: Procedure: Pulsed radiofrequency neuromodulation of the suprascapular nerve only
- PRF three nerves (Active Comparator): Ultrasound guided PRF neuromodulation of suprascapular, axillary nerves, and articular branch of the lateral pectoral nerve
  Interventions: Procedure: Pulsed radiofrequency neuromodulation of the suprascapular, axillary, and articular branch of the lateral pectoral nerves

INTERVENTIONS:
Procedure: Pulsed radiofrequency neuromodulation of the suprascapular nerve only — PRF stimulation of the suprascapular nerve under ultrasound navigation in the notch of the scapula using the Cosman G4 apparatus with the introduction of stimulation: sensory: 50 Hz; 1 ms; up to 0.5 V; motor: 2 Hz; 1 ms; voltage - twice the sensory threshold, but not less than 1V; after introduction of 1 ml of 0.75% ropivacaine, PRF is performed: 42 С, 45V, 2Hz, 20 ms, 1 cycle - 480 sec. Before removing the cannula, local administration of 0.75% ropivacaine 2 ml, dexamethasone 4 mg.
  Under the US navigation, an RF cannula will be placed sequentially at the axillary nerve in the quadrilateral foramen and at the lateral pectoral nerve. After confirmatory sensory and motor stimulation and local administration of 0.75% ropivacaine 1 ml PRF session imitation lasting 480 sec will be carried out. After that local administration of 0.75% ropivacaine 2 ml, dexamethasone 4 mg will follow. The total dose for the entire procedure is ropivacaine 0.75% - 9 ml, dexamethasone 12 mg
  Other Names: PRF one nerve
  Arms: PRF one nerve
Procedure: Pulsed radiofrequency neuromodulation of the suprascapular, axillary, and articular branch of the lateral pectoral nerves — Under ultrasound navigation an RF cannula will be placed sequentially at the suprascapular nerve, at the axillary nerve and at the lateral pectoral nerve. After confirmatory sensory and motor stimulation from RF generator and local administration of 0.75% ropivacaine 1 ml to each nerve, PRF neuromodulation session will be carried out: 42 С, 45V, 2Hz, 20 ms, 1 cycle - 480 sec to each nerve. After that local administration of 0.75% ropivacaine 2 ml, dexamethasone 4 mg will follow to each nerve. The total dose for the entire procedure is ropivacaine 0.75% - 9 ml, dexamethasone 12 mg
  Other Names: PRF three nerves
  Arms: PRF three nerves

SUMMARY:
Pulsed radiofrequency (PRF) neuromodulation / or ablation is an interventional pain management method. Clinical use of PRF for shoulder pain management generally focuses on the suprascapular nerve, what is considered a safe and superior to placebo and physiotherapy. We study the use of the PRF neuromodulation the suprascapular, axillary, and articular branches of the lateral pectoral nerve, as well as the effectiveness of this combined technique compared to the PRF of the suprascapular nerve alone

DETAILED DESCRIPTION:
Background: It's believed that PRf of the suprascapular nerve is a safe and reliable treatment for shoulder pain. But PRF of the suprascapular nerve may be less effective than intra-articular steroid injections (Eyigor et al., 2010). There is also evidence that even test, diagnostic suprascapular nerve blockade in some patients may not give a satisfactory analgesic effect (Sinha et al., 2020). Probably, the unsatisfactory results of PRF suprascapular nerve as a search for a solution force the use of standard thermal RF ablation. (Bone et al., 2013) It is possible to expect a greater clinical effect from the combination of PRF of the three main articular nerves of the suprascapular, axillary and lateral pectoral nerves than from PRF of the suprascapular nerve alone. Nevertheless, having the task of obtaining the maximum effect from PRF, it seems important to maintain a balance between inevitable intervention and excessive intervention, considering that any intervention is associated with the risk of complications.

Methods: The study is planned to include 142 adult patients who are planned to have PRF of the suprascapular nerve due to the presence of chronic shoulder pain.The study is planned as a prospective randomized double-blind controlled trial. According to inclusion / exclusion criteria, written informed consent signing, patients will be randomized in a 1: 1 ratio into two groups: PRF of the suprascapular nerve (n=71) and PRF of the suprascapular, axillary and lateral pectoral nerves (n=71). Patients will be evaluated by a physician 4 weeks and 16 weeks after discharge to receive information on treatment results.

Sample size assessment: To identify differences of 5 points on the SPADI scale at a 5% significance level with 80% power, assuming an expected mean SPADI of 25.5 points and SD - 10.1 according to the study by Korkmaz et al 2010, 64 people will be required for each group. The number 128 was increased to 142 in the sample in order to compensate for observation losses.

ELIGIBILITY:
Inclusion Criteria:

1. Chronic pain (existing for more than three months at the time of examination) in the shoulder associated with the following pathology:

   * rotator cuff injury
   * adhesive capsulitis
   * arthrosis of the shoulder joint
   * arthrosis of the acromioclavicular joint
   * subacromial impingement syndrome
   * a history of arthroscopic surgery
2. Signed informed consent to participate in the study
3. Lack of indications for shoulder surgery
4. Age> 18 years old 5 The positive effect of the test blockade of the suprascapular, axillary and lateral thoracic nerves with a local anesthetic (reduction of the pain level from the baseline according to NRS by at least 50%)

Exclusion Criteria:

1. Rotator cuff calcific tendinopathy
2. infectious arthritis
3. Instability of the shoulder joint
4. cervical radiculopathy
5. contraindications to local anesthetics
6. coagulopathy and anticoagulant therapy
7. pregnancy
8. oncology
9. the impossibility of subjective assessment of the level of pain and function of the joint

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 142 (Estimated)
Dates: Start 2021-08-05 (Actual); Primary Completion 2023-12-30 (Estimated); Study Completion 2024-04-30 (Estimated)

PRIMARY OUTCOMES:
SPADI value | 16 weeks from the time of the procedure
  Scale value Shoulder Pain And Disability Index (SPADI) in points from minimum 0 to maximum 130, where a lower scores means a better outcome

SECONDARY OUTCOMES:
Constant - Murley Shoulder Score | 16 weeks from the time of the procedure
  Scale value Constant - Murley Shoulder Score in points from minimum 0 to maximum 100, where a higher scores means the better of shoulder function.
Recovery in the functionality of the shoulder - DASH value | 16 weeks from the time of the procedure
  Scale value "Disabilities of the Arm, Shoulder and Hand." (DASH) Recovery in the functionality of the shoulder and performing basic activities of daily living from a minimum scale value - 0 (no disability, good functionality) to a maximum - 100 (total disability)
EQ-5D-5L value | 16 weeks from the time of the procedure
  Measuring health-related quality of life according to the EQ-5D-5L questionnaire. Intergroup comparison and deviation from baseline are assessed at 16 weeks from the time of the procedure. Form in the index. Minimum 0 and maximum 1. A higher indicator corresponds to a state of more complete health.

OTHER OUTCOMES:
NSAIDs and opiates needs | 16 weeks from the time of the procedure
  Analyzing in the need for analgesic medication (NSAIDs and opiates)
PRF complications | 16 weeks from the time of the procedure
  Evaluation of complications associated with the implementation of pulsed radiofrequency neuromodulation under ultrasound guidance (neurological, bleeding, hematoma, infection)
Surgical treatment needs | 16 weeks from the time of the procedure
  Evaluation of referral cases for surgical treatment

CONTACTS AND LOCATIONS:
Overall Officials: Konstantin Trukhin, Principal Investigator — Saint Petersburg State University, Russia
Locations (1):
- Saint Petersburg State University, Saint Petersburg, Russia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Korkmaz OK, Capaci K, Eyigor C, Eyigor S. Pulsed radiofrequency versus conventional transcutaneous electrical nerve stimulation in painful shoulder: a prospective, randomized study. Clin Rehabil. 2010 Nov;24(11):1000-8. doi: 10.1177/0269215510371417. Epub 2010 Aug 4. PMID 20685721
- [Result] Eyigor C, Eyigor S, Korkmaz OK, Uyar M. Intra-articular corticosteroid injections versus pulsed radiofrequency in painful shoulder: a prospective, randomized, single-blinded study. Clin J Pain. 2010 Jun;26(5):386-92. doi: 10.1097/AJP.0b013e3181cf5981. PMID 20473045
- [Result] Laumonerie P, Dalmas Y, Tibbo ME, Robert S, Faruch M, Chaynes P, Bonnevialle N, Mansat P. Sensory innervation of the human shoulder joint: the three bridges to break. J Shoulder Elbow Surg. 2020 Dec;29(12):e499-e507. doi: 10.1016/j.jse.2020.07.017. Epub 2020 Jul 23. PMID 32712453